CLINICAL TRIAL: NCT03172780
Title: A Randomized, Double Blind, Three-arm, Parallel, Placebocontrolled, Clinical Study to Evaluate the Bioequivalence Using Clinical Endpoint of Diclofenac Sodium Gel, 1% (Mylan Inc.) to Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% (Novartis Consumer Health, Inc.) in Patients With Osteoarthritis (OA) of the Knee
Brief Title: A Bioequivalence Study Using Clinical Endpoint for Diclofenac Sodium Gel 1% in Osteoarthritis Knee"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Private Limited (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYL-1601N-3002
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Diclofenac Sodium Gel (Experimental): Diclofenac Sodium Gel, 1%
  Interventions: Drug: Diclofenac sodium gel 1%
- Voltaren® Gel (Active Comparator): Voltaren® Gel (Diclofenac Sodium Topical Gel) 1%
  Interventions: Drug: Voltaren® Gel (Diclofenac Sodium Topical Gel) 1%
- Placebo gel (Placebo Comparator): Placebo gel
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Diclofenac sodium gel 1% — Diclofenac Sodium Topical Gel, 1%. 4 gm, 4 times a day for 4 weeks
  Arms: Diclofenac Sodium Gel
Drug: Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% — Diclofenac Sodium Topical Gel, 1%. 4 gm, 4 times a day for 4 weeks
  Arms: Voltaren® Gel
Drug: Placebo gel — Vehicle Gel 4 gm, 4 times a day for 4 weeks
  Arms: Placebo gel

SUMMARY:
This randomized, double-blind, three-arm, placebo controlled, bioequivalence study with clinical endpoint has been designed to establish clinical equivalence and safety of Mylan's diclofenac gel in the symptomatic treatment of osteoarthritis of knee compared to Voltaren® gel and to establish superiority in efficacy of both compared to a placebo (vehicle) gel.

Male or non-pregnant female aged ≥ 35 years with a clinical diagnosis of osteoarthritis of the knee according to the American College of Rheumatology (ACR) criteria

Total study duration for the clinical part will be around 56 days that includes screening period of 28 days and treatment period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis knee as per American College of Rheumatology (ACR) criteria
* Evidence of OA with Kellgren-Lawrence grade 1-3 disease.
* After discontinuing all pain medications, had at least moderate pain on movement (POM) for target knee
* After discontinuing all pain medications for at least 7 days has a baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC Likert (version 3.1)) pain subscale of ≥ 9 immediately prior to randomization.
* Able to tolerate rescue medication with acetaminophen
* Subjects who can read and understand WOMAC pain sub scale

Exclusion Criteria:

* Pregnancy, lactation
* OA of Kellgren-Lawrence grade 4
* OA pain in the contralateral knee requiring medication (OTC or prescription)
* History of OA of either Hip or Hands
* History of secondary OA (e.g. congenital, traumatic, gouty arthritis), rheumatoid arthritis
* History of chronic inflammatory disease (e.g., colitis) or fibromyalgia
* History of Drugs or Alcohol abuse within the previous year
* Symptomatic peripheral vascular disease of the study leg
* Any musculoskeletal condition
* Skin disease at the application site
* Active asthma requiring periodic treatment with systemic steroids
* Known history of positive HIV, hepatitis C virus, or HBsAg
* Uncontrolled hypertension
* History of myocardial infarction, thrombotic events, stroke etc.
* Allergy to aspirin, nonsteroidal anti-inflammatory drugs (NSAID) or acetaminophen (paracetamol).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- India (32):
  - Yashoda Hospital - Malakpet, Hyderabad, Andhra Pradesh
  - Yashoda Hospital -Secunderabad, Secunderabad, Andhra Pradesh
  - Yashoda Hospital -Somajiguda, Somajiguda, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Riddhi Medical Nursing Home, Ahmedabad, Gujarat
  - Rathi Hospital, Ahmedabad, Gujarat
  - Sanjivani Superspeciality Hospital Pvt. Ltd, Ahmedabad, Gujarat
  - B.J Medical College & Civil Hospital, Ahmedabad, Gujarat
  - GMERS Medical College & Civil Hospital, Ahmedabad, Gujarat
  - Medistar Multispeciality Hospital, Himmatnagar, Gujarat
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - SSG Hospital and Medical College, Vadodara, Gujarat
  - Anand Multispeciality Hospital, Vadodara, Gujarat
  - Parul Sevashram Hospital, Vadodara, Gujarat
  - Omega Hospital, Mangalore, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - Sree Narayana Institute of Medical Science, Ernākulam, Kerala
  - Sir J. J. Group of Hospital and Grant Government Hospital, Mumbai, Maharashtra
  - Lokmanya Tilak Municipal Medical College & General Hospital, Mumbai, Maharashtra
  - Government Medical College and Hospital, Nagpur, Maharashtra
  - Jasleen Hospital, Nagpur, Maharashtra
  - Institute of Medical sciences and Lata Mangeshkar, Nagpur, Maharashtra
  - Supe Heart and Diabetes Hospital & Research Centre, Nashik, Maharashtra
  - BJ medical college & Sassoon General Hospital, Pune, Maharashtra
  - Sancheti Institute for Orthopedics & Rehabilitation, Pune, Maharashtra
  - BhaktiVedanta Hospital and Research Institute, Thane, Maharashtra
  - IMS and SUM Hospital, Bhubaneshwar, Odisha
  - Govt Stanley Medical College & Hospital, Chennai, Tamil Nadu
  - M.V. Hospital & Research Centre, Lucknow, Uttar Pradesh
  - Ajanta Research Centre, Lucknow, Uttar Pradesh
  - OM surgical Centre and Maternity Home, Varanasi, Uttar Pradesh
  - Institute of Post Graduate Medical Education and Research (IPGMER), Department of Orthopaedics, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diclofenac Sodium Gel | Voltaren® Gel | Placebo Gel
Started | 406 | 409 | 405
Completed | 388 | 389 | 389
Not Completed | 18 | 20 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium Gel | Voltaren® Gel | Placebo Gel | Total
Number analyzed (Participants) | 406 | 409 | 405 | 1220
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (9.51) | 53.4 (9.40) | 53.6 (10.15) | 53.4 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 288 | 273 | 836
  Male | 131 | 121 | 132 | 384
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Not Hispanic or Latino | 406 | 409 | 405 | 1220
Region of Enrollment [Number; unit: participants]
  India | 406 | 409 | 405 | 1220
WOMAC Pain subscale score for target knee [Mean (Standard Deviation); unit: units on a scale] — Western Ontario and McMaster Universities Osteoarthritis Index WOMAC pain subscale score (pain score = minimum 0 to maximum 20), was determined by the sum of subject's responses to five questions (S1-S5) using a 5-point Likert scale (i.e., 'none'=0; 'mild'=1, 'moderate'=2; 'severe'=3; 'extreme'=4). Higher values represent worse outcome.
  'How much pain do you have' when 'Walking on a flat surface' (S1), 'Going up or down stairs' (S2), 'at night while in bed' (S3), 'Sitting or lying' (S4), 'Standing upright' (S5)].
  units on a scale | 12.4 (2.15) | 12.5 (2.16) | 12.4 (2.05) | 12.4 (2.12)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Total WOMAC Pain Subscale Score
Description: Mean change in the total WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) pain subscale score for the target knee was compared to determine the clinical equivalence of Test Drug (Diclofenac sodium gel of 1% of Mylan Inc.) with the Reference Listed Drug (RLD) (Voltaren® Gel 1% of Novartis Consumer Health, Inc.) Measure Description: Western Ontario and McMaster Universities Osteoarthritis Index WOMAC pain subscale score (pain score = min 0 to max 20), was determined by the sum of subject's responses to five questions (S1-S5) using a 5-point Likert scale (i.e., 'none'=0; 'mild'=1, 'moderate'=2; 'severe'=3; 'extreme'=4). Higher values represent worse outcome.
  'How much pain do you have' when 'Walking on a flat surface' (S1), 'Going up or down stairs' (S2), 'at night while in bed' (S3), 'Sitting or lying' (S4), 'Standing upright' (S5)].
  The timepoints considered for the primary outcomes include baseline and week 4.
Time Frame: From baseline to week 4
Population: The PP Population was used for analysis of clinical equivalence between Mylan's Diclofenac gel and Voltaren gel. The primary outcome tested in this population was the equivalence of Mylan's Diclofenac sodium gel (1%) verses the Voltaren gel (1%) and thus only Diclofenac Sodium Gel and Voltaren Gel arms are present here. The placebo arm is presented for the superiority analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diclofenac Sodium Gel | Voltaren® Gel
Number analyzed (Participants) | 318 | 330
score on a scale | -4.3 (2.64) | -4.6 (2.64)

2. Primary Outcome: Change From Baseline in WOMAC Pain Subscale Score
Description: Mean change in the total WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) pain subscale score for the target knee was compared to determine the superiority of the Test Drug and Reference Listed Drug (RLD) over placebo.
  Measure Description: Western Ontario and McMaster Universities Osteoarthritis Index WOMAC pain subscale score (pain score = min 0 to max 20), was determined by the sum of subject's responses to five questions (S1-S5) using a 5-point Likert scale (i.e., 'none'=0; 'mild'=1, 'moderate'=2; 'severe'=3; 'extreme'=4). Higher values represent worse outcome.
  'How much pain do you have' when 'Walking on a flat surface' (S1), 'Going up or down stairs' (S2), 'at night while in bed' (S3), 'Sitting or lying' (S4), 'Standing upright' (S5)].
  The timepoints considered for the primary outcomes include baseline and week 4.
Time Frame: 4 weeks
Population: The mITT Population was used for analysis of superiority of Mylan's Diclofenac gel and Voltaren gel over placebo. The primary outcome tested in this population was the superiority of Mylan's Diclofenac sodium gel (1%) and the Voltaren gel (1%) over placebo and thus all the three arms are presented here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diclofenac Sodium Gel | Voltaren® Gel | Placebo Gel
Number analyzed (Participants) | 386 | 402 | 396
score on a scale | -4.2 (2.84) | -4.4 (2.74) | -3.2 (3.46)

ADVERSE EVENTS:
Time Frame: The reporting period for TEAEs started after the informed consent through day 28 after the last application of investigational product, a total of approximately 12 weeks.
Description: The safety analysis was performed based on safety population that includes all patients who were treated with at least one application of the investigational product. The total number of patients included in this population were 1203 (398 for Mylan's Diclofenac gel, 405 for Voltaren gel and 400 for placebo).
Arm/Group | Diclofenac Sodium Gel | Voltaren® Gel | Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/398 | 1/405 | 0/400
Serious Adverse Events (participants affected / at risk) | 0/398 | 1/405 | 0/400
Other Adverse Events (participants affected / at risk) | 11/398 | 19/405 | 20/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Gel (N=398) | Voltaren® Gel (N=405) | Placebo Gel (N=400)
Completed Suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Gel (N=398) | Voltaren® Gel (N=405) | Placebo Gel (N=400)
Headache (Nervous system disorders) | 4 (5) | 9 (12) | 11 (14)
Pyrexia (General disorders) | 6 (6) | 6 (9) | 9 (11)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03172780/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03172780/SAP_001.pdf